CLINICAL TRIAL: NCT02688426
Title: Effects Acute of the Low-level Laser Therapy on Functional Capacity on Patients With Coronary Artery Bypass Surgery : A Randomized, Controlled Clinical Trail
Brief Title: Effects of the Low-level Laser Therapy on Functional Capacity of the Patients With Coronary Artery Bypass Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, Clinical Research, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LLLT-CABG-2016/1
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0J LLLT (Sham Comparator): The sham treatment is performed in the same way as treatment with LBP, however, with the apparatus switched off
  Interventions: Device: Sham Low-Level Laser Therapy (Sham LLLT); Device: 6J Low-Level Laser Therapy (6J LLLT)
- 6J LLLT (Experimental): The Laser radiation will be made with 6J by spot.
  Interventions: Device: Sham Low-Level Laser Therapy (Sham LLLT); Device: 6J Low-Level Laser Therapy (6J LLLT)

INTERVENTIONS:
Device: Sham Low-Level Laser Therapy (Sham LLLT) — perform with the machine off
  Other Names: Sham LLLT
Device: 6J Low-Level Laser Therapy (6J LLLT) — irradiation will be perform with 6J
  Other Names: 6J

SUMMARY:
The low-level laser therapy (LLLT) has been used in many inflammatory disorders.

More recently the LLLT was associated with an improvement in the muscle strength, endurance and functional capacity.But, these effects were described only in health or athletic individuals. In this randomized and controlled clinical trails, the investigators will study the effects of LLLT on functional capacity of the patients with Coronary artery bypass surgery.

DETAILED DESCRIPTION:
This study will be conducing in a large hospital that is reference in Coronary artery bypass surgery. 15 patients will be randomized for placebo or low-level laser therapy (LLLT). The functional capacity will be test by test six-minute walk test before and after de LLLT. Moreover the application of LBP or placebo will be followed by assessments of muscle damage and oxidative stress. One-week interval between the LLLT will gave to reduce the influence between the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the postoperative period of elective CABG referred for cardiac rehabilitation, which are the 15th and 30th days after surgery without ischemic changes and / or complex arrhythmias on the electrocardiogram, between 40 and 75 years of age who have performed the first surgery.

Exclusion Criteria:

* Patients with decompensated heart failure; presence of any comorbidity such as: unstable angina; associated neurological disease; moderate respiratory illness to severe pre-diagnosed by the attending physician; active infectious disease or fever; disabling peripheral vascular disease; unstable ventricular arrhythmias; diabetes mellitus; use of cardiac pacemaker, musculoskeletal disease that limits physical activity, patients with a BMI ≥30.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | up to 2 weeks

SECONDARY OUTCOMES:
Muscle damage | up to 2 weeks
  The damage to DNA is analyzed by electrophoresis single (comet technique), where cells are counted by microscopy.
Oxidative stress | up to 2 weeks
  Oxidative stress will be used a measure of tissue damage, the protein oxidation (method of carbonyls) and two defense measures, an enzyme superoxide dismutase and total antioxidant capacity. Oxidative damage (nmol / mg) of protein carbonylation was determined according to the method proposed by Levine & Stadtman, 1990, using whole blood. The enzymatic activity of SOD (SOD / mg protein) was determined by the inhibition of autooxidation of adrenaline measured spectrophotometrically (480nm) under Bannister and Calabrese (1987).

CONTACTS AND LOCATIONS:
Locations (1):
- Rodrigo Della Méa Plentz, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stein C, Fernandes RO, Miozzo AP, Coronel CC, Baroni BM, Bello-Klein A, Plentz RDM. Acute Effects of Low-Level Laser Therapy on Patients' Functional Capacity in the Postoperative Period of Coronary Artery Bypass Graft Surgery: A Randomized, Crossover, Placebo-Controlled Trial. Photomed Laser Surg. 2018 Mar;36(3):122-129. doi: 10.1089/pho.2017.4270. Epub 2018 Feb 21. PMID 29466116